CLINICAL TRIAL: NCT03601390
Title: Combining Fluorodeoxyglucose-Positron Emission Tomography/Computed Tomography and Plasma EBV DNA to Evaluate the Hazard of Progression in the Follow-up of Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Combining PET/CT and EBV DNA to Evaluate the Hazard of Progression in the Follow-up of Locally Advanced NPC
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, prof. Haiqiang Mai, Sun Yat-sen University
Other Study IDs: Post-treament PET/CT in NPC
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: PET/CT; EBV DNA; predicting predicting
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PET/CT and EBV DNA: Patients receiving chemoradiotherapy will receive a dedicated FDG PET/CT protocol 12 weeks after the end of IMRT (primary endpoint).Plasma EBV DNA test will be performed 4, 12, 24 weeks after the end of IMRT. In patients with negative PET/CT results, 2 follow-up visits are required to complement nasopharyngoscope examination and plasma EBV DNA test in the frist year. All patients will undergo annual PET/CT or traditional follow-up examination and plasma EBV DNA test 1 year after completing chemoradiation unless recurrent/residual disease is histopathologically-confirmed.
  Interventions: Device: PET/CT and EBV DNA

INTERVENTIONS:
Device: PET/CT and EBV DNA — PET/CT and EBV DNA will be proformed after the IMRT treatment

SUMMARY:
PET/CT and EBV DNA are important in diagnosis of NPC. We consider that combining post-treament PET/CT and plasma EBV DNA may be effective in evaluating the hazard of progression in the follow-up of Locally Advanced Nasopharyngeal Carcinoma. Hence we establish this prospective cohort study.

DETAILED DESCRIPTION:
Newly-diagnosed patients with stage III or IV non-metastatic Nasopharyngeal Carcinoma (AJCC 7th) will be recruited. All subjects receiving chemoradiotherapy will undergo a baseline integrated [18F]fluoro-2-deoxy-D-glucose (FDG) positron emission tomography/computed tomography (PET/CT) scan or traditional follow-up examination and plasma EBV DNA test before the start of chemoradiotherapy.

Patients receiving IMRT treatment will receive a dedicated FDG PET/CT protocol 12 weeks after the end of chemoradiotherapy (primary endpoint).Plasma EBV DNA test will be performed 4, 12, 24 weeks after the end of IMRT treatment. In patients with negative PET/CT results, 2 follow-up visits are required to complement nasopharyngoscope examination and plasma EBV DNA test in the frist year. All patients will undergo annual PET/CT or traditional follow-up examination and plasma EBV DNA test 1 year after completing chemoradiation unless recurrent/residual disease is histopathologically-confirmed.

Patients with a PET/CT result suspecting for residual/recurrent/metastatic tumor must have pathological and/or clinical evidence of tumor existence before salvage therapy is started.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and given written informed consent.
* Aged between 18-65, male/female.
* Staged III or IV (AJCC 7th) NPC patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma (including differentiated type and undifferentiated type, WHO II and III).
* Received induction chemotherapy and/or concurrent chemoradiotherapy.
* ECOG scale 0-1.
* Fertile women should practice contraception during the study period.
* HGB ≥90g/L ,WBC ≥4*109/L , PLT ≥100*109/L,
* With normal liver function test (ALT and AST ≤2.5*ULN, TBil ≤2.0*ULN)
* With normal renal function test (serum creatinine ≤1.5*ULN)

Exclusion Criteria:

* Women in pregnancy or lactation
* Prior malignancy except adequately treated basal cell, squamous cell skin cancer, or cervical cancer in situ.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.
* Already involved in other clinical trial.
* Mental disorder, civil disability, limited capacity for civil conduct.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NPC patients after induction chemotherapy and concurrent chemoradiotherapy or concurrent chemoradiotherapy alone
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of FDG PET/CT | 12 weeks after IMRT treatment
  The negative predictive value (NPV) of FDG PET/CT for detecting tumor existence

SECONDARY OUTCOMES:
Negative predictive value (NPV) of EBV DNA | 2-year
  Negative predictive value (NPV) of EBV DNA for detecting tumor existence
PFS | 2-year
  progression free survival after radical treatment
Negative predictive value (NPV) of combined EBV DNA and FDG PET/CT | 2-year
  Negative predictive value (NPV) of combined EBV DNA and FDG PET/CT for detecting tumor existence
OS | 2-year
  overall survival after radical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, Dr, Study Chair — Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van den Wyngaert T, Helsen N, Carp L, Hakim S, Martens MJ, Hutsebaut I, Debruyne PR, Maes ALM, van Dinther J, Van Laer CG, Hoekstra OS, De Bree R, Meersschout SAE, Lenssen O, Vermorken JB, Van den Weyngaert D, Stroobants S; ECLYPS investigators. Fluorodeoxyglucose-Positron Emission Tomography/Computed Tomography After Concurrent Chemoradiotherapy in Locally Advanced Head-and-Neck Squamous Cell Cancer: The ECLYPS Study. J Clin Oncol. 2017 Oct 20;35(30):3458-3464. doi: 10.1200/JCO.2017.73.5845. Epub 2017 Aug 30. PMID 28854069
- [Background] Marcus C, Ciarallo A, Tahari AK, Mena E, Koch W, Wahl RL, Kiess AP, Kang H, Subramaniam RM. Head and neck PET/CT: therapy response interpretation criteria (Hopkins Criteria)-interreader reliability, accuracy, and survival outcomes. J Nucl Med. 2014 Sep;55(9):1411-6. doi: 10.2967/jnumed.113.136796. Epub 2014 Jun 19. PMID 24947059
- [Background] Dibble EH, Alvarez AC, Truong MT, Mercier G, Cook EF, Subramaniam RM. 18F-FDG metabolic tumor volume and total glycolytic activity of oral cavity and oropharyngeal squamous cell cancer: adding value to clinical staging. J Nucl Med. 2012 May;53(5):709-15. doi: 10.2967/jnumed.111.099531. Epub 2012 Apr 9. PMID 22492732
- [Background] Imsande HM, Davison JM, Truong MT, Devaiah AK, Mercier GA, Ozonoff AJ, Subramaniam RM. Use of 18F-FDG PET/CT as a predictive biomarker of outcome in patients with head-and-neck non-squamous cell carcinoma. AJR Am J Roentgenol. 2011 Oct;197(4):976-80. doi: 10.2214/AJR.10.4884. PMID 21940588
- [Background] Chen QY, Guo SY, Tang LQ, Lu TY, Chen BL, Zhong QY, Zou MS, Tang QN, Chen WH, Guo SS, Liu LT, Li Y, Guo L, Mo HY, Sun R, Luo DH, Zhao C, Cao KJ, Qian CN, Guo X, Zeng MS, Mai HQ. Combination of Tumor Volume and Epstein-Barr Virus DNA Improved Prognostic Stratification of Stage II Nasopharyngeal Carcinoma in the Intensity Modulated Radiotherapy Era: A Large-Scale Cohort Study. Cancer Res Treat. 2018 Jul;50(3):861-871. doi: 10.4143/crt.2017.237. Epub 2017 Sep 13. PMID 28903550
- [Background] Chen QY, Tang QN, Tang LQ, Chen WH, Guo SS, Liu LT, Li CF, Li Y, Liang YJ, Sun XS, Guo L, Mo HY, Sun R, Luo DH, Fan YY, He Y, Chen MY, Cao KJ, Qian CN, Guo X, Mai HQ. Pretreatment Serum Amyloid A and C-reactive Protein Comparing with Epstein-Barr Virus DNA as Prognostic Indicators in Patients with Nasopharyngeal Carcinoma: A Prospective Study. Cancer Res Treat. 2018 Jul;50(3):701-711. doi: 10.4143/crt.2017.180. Epub 2017 Jul 14. PMID 28707462
- [Background] Davison JM, Ozonoff A, Imsande HM, Grillone GA, Subramaniam RM. Squamous cell carcinoma of the palatine tonsils: FDG standardized uptake value ratio as a biomarker to differentiate tonsillar carcinoma from physiologic uptake. Radiology. 2010 May;255(2):578-85. doi: 10.1148/radiol.10091479. PMID 20413767
- [Background] Paidpally V, Tahari AK, Lam S, Alluri K, Marur S, Koch W, Wahl RL, Subramaniam RM. Addition of 18F-FDG PET/CT to clinical assessment predicts overall survival in HNSCC: a retrospective analysis with follow-up for 12 years. J Nucl Med. 2013 Dec;54(12):2039-45. doi: 10.2967/jnumed.113.121285. Epub 2013 Oct 7. PMID 24101687
- [Background] Sherriff JM, Ogunremi B, Colley S, Sanghera P, Hartley A. The role of positron emission tomography/CT imaging in head and neck cancer patients after radical chemoradiotherapy. Br J Radiol. 2012 Nov;85(1019):e1120-6. doi: 10.1259/bjr/20976707. Epub 2012 Jun 27. PMID 22744325
- [Background] Wong RJ. Current status of FDG-PET for head and neck cancer. J Surg Oncol. 2008 Jun 15;97(8):649-52. doi: 10.1002/jso.21018. PMID 18493944